CLINICAL TRIAL: NCT00017823
Title: The Acupressure Study
Brief Title: Acupressure to Treat Nausea and Vomiting in HIV/AIDS Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 9941
Record Dates: First submitted 2001-06-13; First posted 2001-06-14 (Estimated); Last update posted 2010-04-21 (Estimated); Status verified 2001-04

CONDITIONS: HIV Infections
Keywords: complementary therapies; Acupressure; HIV Infections; Nausea; Vomiting
MeSH Terms: conditions — HIV Infections; Nausea; Vomiting | interventions — Acupressure

INTERVENTIONS:
Procedure: Acupressure

SUMMARY:
The purpose of this study is to see whether acupressure (acupuncture using pressure applied by the hands instead of needles) can help nausea and vomiting in persons with HIV/AIDS.

DETAILED DESCRIPTION:
This is a Phase I trial (a study to evaluate effectiveness in a small number of patients). Patients will get 4 acupressure treatments and will wear acupressure wristbands for 1 week. Patients will write down all drugs they take and will make a note of when they get nausea and vomiting. They also will give written answers to different questions. No drugs will be given as part of this study. Patients will be paid for participating.

ELIGIBILITY:
Inclusion Criteria:

* Are HIV-positive.
* Have nausea and/or vomiting an average of 2 times per day for at least 1 week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia Univ School of Nursing / Center for AIDS Research, New York, New York, United States